CLINICAL TRIAL: NCT06327048
Title: Application of Cognitive Training Based on Remind Strategy in Glioma Patients With Cognitive Impairment
Brief Title: Application of Cognitive Training Based on the Remind Strategy in Glioma Patients With Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: YuanYuan Ma (Other)
Responsible Party: Sponsor-Investigator, YuanYuan Ma, supervisor nurse, LanZhou University
Organization: LanZhou University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: LZUHLXY20230110
Record Dates: First submitted 2024-02-29; First posted 2024-03-25 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2024-10

CONDITIONS: Glioma
Keywords: cognitive training; cognitive impairment; Quality of Life
MeSH Terms: conditions — Glioma; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Non-randomized intervention study
Who Masked: Outcomes Assessor
Masking Description: Blind the evaluator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Routine rehabilitation nursing
- Intervention group (Experimental): On the basis of routine rehabilitation nursing, individual cognitive rehabilitation training based on Remind strategy was given
  Interventions: Other: Individual cognitive rehabilitation training based on Remind strategy was given

INTERVENTIONS:
Other: Individual cognitive rehabilitation training based on Remind strategy was given — This training educates and learns patients from the aspects of assessment of cognitive function and strategic compensation for the impact of cognitive impairment on patients, and then conducts attention, memory and executive function training and attention retraining based on patients' cognitive function to improve patients' cognitive function
  Arms: Intervention group

SUMMARY:
The purpose of this study is to form an interdisciplinary team to dynamically evaluate patient cognitive outcomes and develop an individualized cognitive training program for Chinese brain tumor patients

DETAILED DESCRIPTION:
Adult patients diagnosed with glioma who meet the inclusion criteria will be enrolled in this study. Patients admitted to Neurosurgery Ward 1 will be assigned to the intervention group, while those admitted to Neurosurgery Ward 2，ward 3 and Ward 4 will serve as the control group. The intervention group will receive cognitive rehabilitation training based on the Remind strategy in addition to standard rehabilitation care, whereas the control group will receive only standard rehabilitation care. Assessment of patients' cognitive function, quality of life, psychological status, and the effectiveness of cognitive training intervention will be conducted on the first day of admission, before intervention, at the end of the 4-week and 12-week intervention .

ELIGIBILITY:
Inclusion Criteria:

1. Conforming to the diagnostic criteria outlined in the "Chinese Clinical Guidelines for Diagnosis and Treatment of Central Nervous System Gliomas (2015)" ;
2. Patients diagnosed with brain gliomas through histopathological and/or cytological examination;
3. MoCA (Montreal Cognitive Assessment) score ≤ 26;
4. Karnofsky Performance Status (KPS) score ≥ 60, with no history of past illnesses;
5. Age ≥ 18 years;
6. Clear consciousness;
7. Willingness to participate and signed informed consent form.

Exclusion Criteria:

1. Diagnosed with neurological or psychiatric disorders within the past two years;
2. Impaired consciousness;
3. Accompanied by severe complications such as infections;
4. Nursing Delirium Screening Checklist (Nu-DESC) score ≥ 2;
5. Patients with changes in condition or requiring repeat surgery;
6. Patients with multiple intracranial tumors;
7. Inability to effectively complete the questionnaire or withdrawal during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2024-01-21 (Actual); Primary Completion 2025-01-12 (Actual); Study Completion 2025-01-12 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment(MoCA) | The day after admission, 7 days after surgery (baseline), at 4-week and 12-week of intervention.
  The Montreal Cognitive Assessment (MoCA) is commonly used to assess cognitive function, typically taking about 15 minutes to complete. It has a total score of 30 points, with a score of ≥26 considered normal. Lower scores indicate more severe cognitive impairment. MoCA is advantageous due to its ease of administration, short duration, and high reliability and validity.

SECONDARY OUTCOMES:
The European Organization for Research and Treatment of Cancer core Quality of Life Questionnaire (EORTC QLQ-C30) | The day after admission, 7 days after surgery (baseline), at 4-week and 12-week of intervention.
  The European Organization for Research and Treatment of Cancer core Quality of Life Questionnaire (EORTC QLQ-C30) includes five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea and vomiting), a global health and QoL scale, as well as individual items to assess other symptoms commonly experienced by cancer patients (such as dyspnea, appetite loss, sleep disturbance, constipation, and diarrhea), and the perceived economic impact of the disease and treatment. All items are scored using a 4-point Likert scale (1: 'not at all'; to 4: 'very much'), except for two items in the global health/QoL scale which use a modified 7-point linear analog scale. Higher scores indicate poorer quality of life.
The EORTC QLQ-Brain Neoplasms 20(EORTC QLQ-BN20) | The day after admission, 7 days after surgery (baseline), at 4-week and 12-week of intervention.
  The EORTC QLQ-Brain Neoplasms 20(EORTC QLQ-BN20) is a tool specifically designed to assess the quality of life of patients with brain tumors. The instrument consists of four multi-item scales covering: future uncertainty; visual disorders; motor dysfunction; communication deficit. Additionally, seven individual items assess headache, seizures, drowsiness, hair loss, itching, weakness of legs, and bladder control. All items and scores are evaluated on a scale of 0-100, with higher scores reflecting more severe symptoms.
Self-Rating Anxiety Scale(SAS) | The day after admission, 7 days after surgery (baseline), at 4-week and 12-week of intervention.
  The Self-Rating Anxiety Scale (SAS) is used to assess the subjective feelings of anxiety patients. The scale consists of 20 items aimed at quantifying the severity of anxiety-related symptoms experienced by patients. It is divided into four levels on a Likert four-point scale: None or rarely, Sometimes, Often, and Always. Scores range from 20 to 80, with 20-44 considered normal, 45-59 indicating mild to moderate anxiety levels, 60-74 indicating severe anxiety levels, and extreme anxiety levels falling between 75 and 80.
Self-Rating Depression Scale(SDS) | The day after admission, 7 days after surgery (baseline), at 4-week and 12-week of intervention.
  The Self-Rating Depression Scale (SDS) is used to assess an individual's subjective feelings of depression. The scale consists of 20 items rated on a Likert four-point scale: None or rarely, Sometimes, Often, and Always. Higher scores indicate higher levels of depression in the individual.
Modified Barthel Index(MBI) | The day after admission, 7 days after surgery (baseline), at 4-week and 12-week of intervention.
  The Modified Barthel Index (MBI) is widely used in clinical practice to assess activities of daily living (ADL). It reflects patients' ability to perform self-care activities such as dressing, feeding, personal hygiene, as well as mobility activities such as sitting, standing, and walking. This scale is straightforward, easy to administer, and has good reliability and validity.

CONTACTS AND LOCATIONS:
Overall Officials: peifen ma, Master, Study Director — Lanzhou University Second Hospital
Locations (1):
- Yuanyuanma, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No
The research data is being preserved by the research team and will be presented in the published paper after the study is completed.